CLINICAL TRIAL: NCT01893580
Title: Perioperative Rehabilitation in Operation for Lung Cancer
Acronym: PROLUCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low recruiment rate, the study design is chanced to a feasibility study
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Centre for Integrated Rehabilitation of Cancer patients, CIRE, Denmark (Unknown); Danish Cancer Society (Other); Novo Nordisk A/S (Industry); University of Copenhagen (Other); Copenhagen Centre for Cancer and Health, Denmark. (Unknown)
Responsible Party: Principal Investigator, Jesper Holst Pedersen, MD, DrMSci, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROLUCA; 2007-58-0015 (Registry Identifier: Danish Data Protection Agency)
Record Dates: First submitted 2013-06-20; First posted 2013-07-09 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: Cancer; Rehabilitation; Exercise; Lung cancer; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1. Experimental (Experimental): Home-based exercise pre surgery and postoperative exercise in a team initiated two weeks after surgery.
  Interventions: Behavioral: Experimental: 1. Experimental
- 2. Experimental (Experimental): Home-based exercise pre surgery and postoperative exercise in a team initiated six weeks after surgery.
  Interventions: Behavioral: Experimental: 2. Experimental
- 3. Experimental (Experimental): Exercise in a team initiated two weeks after surgery.
  Interventions: Behavioral: Experimental: 3. Experimental
- 4. Usual care (Other): Exercise in a team initiated six weeks after surgery.
  Interventions: Behavioral: Other: 4. Usual care

INTERVENTIONS:
Behavioral: Experimental: 1. Experimental — Home-based exercise pre surgery and postoperative exercise in a team initiated two weeks after surgery. Intervention consists of:
  1. Preoperative home-based exercise program - cardiovascular exercise of moderate-vigorous intensity for at least 30 minutes every day until surgery.
  2. Postoperative rehabilitation: A supervised 12-week rehabilitation program containing 24 group-based exercise sessions, three individual counseling sessions and smoking cessation, nutritional counseling or patient education, this is offered too.The cardiorespiratory intensity is at ~50-60% of individual HRmax for the first four weeks and increases to moderate-high intensity at ~70-90% of individually determined HRmax. The intensity of the strength exercise program is at ~60-80% of 1 RM.
  Other Names: Preoperative and early postoperative rehabilitation
  Arms: 1. Experimental
Behavioral: Experimental: 2. Experimental — Home-based exercise pre surgery and postoperative exercise in a team initiated six weeks after surgery. Intervention consists of:
  1. Preoperative home-based exercise program - cardiovascular exercise of moderate-vigorous intensity for at least 30 minutes every day until surgery.
  2. Postoperative rehabilitation: A supervised 12-week rehabilitation program containing 24 group-based exercise sessions, three individual counseling sessions and smoking cessation, nutritional counseling or patient education, this is offered too.The cardiorespiratory intensity is at ~50-60% of individual HRmax for the first four weeks and increases to moderate-high intensity at ~70-90% of individually determined HRmax. The intensity of the strength exercise program is at ~60-80% of 1 RM.
  Other Names: Preoperative and late postoperative rehabilitation
  Arms: 2. Experimental
Behavioral: Experimental: 3. Experimental — Early postoperative exercise in a team initiated two weeks after surgery. Intervention consists of:
  Postoperative rehabilitation: A supervised 12-week rehabilitation program containing 24 group-based exercise sessions, three individual counseling sessions and smoking cessation, nutritional counseling or patient education, this is offered too.The cardiorespiratory intensity is at ~50-60% of individual HRmax for the first four weeks and increases to moderate-high intensity at ~70-90% of individually determined HRmax. The intensity of the strength exercise program is at ~60-80% of 1 RM.
  Other Names: Early postoperative rehabilitation alone
  Arms: 3. Experimental
Behavioral: Other: 4. Usual care — Exercise in a team initiated six weeks after surgery consisting of a supervised 12-week rehabilitation program containing 24 group-based exercise sessions, three individual counseling sessions, and three group-based lessons in health-promoting behavior. If the participants have special needs in terms of smoking cessation, nutritional counseling or patient education, this is offered too.
  The cardiorespiratory intensity is at ~50-60% of individual HRmax for the first four weeks. The next eight weeks the intensity increases to moderate-high intensity at ~70-90% of individually determined HRmax. The intensity of the strength exercise program is at ~60-80% of 1 RM.
  Other Names: Usual care
  Arms: 4. Usual care

SUMMARY:
Background: Improved surgical techniques combined with effective adjuvant chemotherapy, has led to a better survival in individuals with NSCLC. The treatment of NSCLC and other cancer diseases are after all still complex and potentially lethal.

Study aim: The rationale for the study PROLUCA is to identify the optimal timing of exercise to improve recovery after surgery in patients operated for lunge cancer with focus on physical capacity and quality of life.

Who can participate? Patients above 18 years and diagnosed with lung cancer and referred for operation. Participation in this study is not possible if the participants by a doctor are advised not to do strenuous exercise.

What does the study involve? The intervention consists of a combination of (1) exercise before surgery and (2) exercise after surgery for lung cancer.

1. Exercise before surgery is a home-based exercise program is individually designed and must be performed for at least 30 minutes every day until surgery. The home-based exercise program varies in length due to number of days until surgery, and the intention is not exceed 14 days.
2. The exercise initiated two weeks and 6 weeks after surgery consists of a 12 weeks rehabilitation program and three individual counseling sessions. Special needs in terms of smoking cessation, nutritional counseling or patient education, this is also offered. The exercise consists of individually prepared supervised strength - and fitness exercise in a team, two sessions of 60 minutes/week.

What interventions will be compared? A home-based post-operative exercise program, combined with exercise initiated two weeks after surgery, will be compared with usual care (exercise initiated six weeks after surgery).

Will all participants receive the same treatment?

By draw it is decided which of the 4 groups the participants will attend to in the study:

* Group 1: Home-based exercise before surgery and rehabilitation initiated as early as two weeks after surgery
* Group 2: Home-based exercise before surgery and rehabilitation initiated six weeks after surgery
* Group 3: Rehabilitation initiated as early as two weeks after surgery
* Group 4: Rehabilitation initiated six weeks after surgery (Usual practice as control group) What are the possible benefits and risks of participating? There are no risks or side- effects of participating other than muscle soreness and exercise is beneficial when it comes to recover from an operation from lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Performance status 0-2 (WHO)
* Living in the City of Copenhagen or surrounding Municipalities
* Ability to read and understand Danish
* Approval by primary surgeon

Exclusion Criteria:

* Presence of metastatic disease or surgical inoperability
* Diagnosis of Lung Cancer not verified by histological diagnosis
* Cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen uptake (VO2peak) | VO2peak is assessed at baseline, the day before surgery, post-intervention (14/18 weeks after surgery), six months after surgery, and one year after surgery.
  VO2peak is evaluated by an incremental test using an electromagnetically braked cycle ergometer (Lode Corival Ergometer©). Inspired and expired gases are analyzed breath-by-breath by a metabolic cart (JAEGER MasterScreen CPX©). Subjects begin pedaling at seven watts and resistance increases after a predefined 10 watts ramp protocol until exhaustion or a symptom-limited VO2peak is achieved (pain, dizziness, anxiety etc.).

SECONDARY OUTCOMES:
Six minute walk distance (6MWD) | baseline, the day before surgery, pre-intervention (2/6 weeks after surgery), post-intervention (14/18 weeks after surgery), six months after surgery, and one year after surgery.
Patient reported outcomes (PROs) | Baseline, the day before surgery, pre-intervention (2/6 weeks after surgery), post-intervention (14/18 weeks after surgery), six months after surgery, and one year after surgery.
  PROs will include health related quality of life, symptoms and side-effects, anxiety and depression, well-being, distress, lifestyle, sickness absence, work status, and social support.
Pulmonary function | Baseline, the day before surgery, post-intervention (14/18 weeks after surgery), six months after surgery, and one year after surgery.
  forced expiratory volume at one second

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Holst Pedersen, MD, DrMSci, Study Chair — Department of Cardiothoracic Surgery RT; Jette Vibe-Petersen, MD, Study Director — Copenhagen Centre for Cancer and Health; Maja Schick Sommer, MHS, Principal Investigator — Copenhagen Centre for Cancer and Health
Locations (1):
- Copenhagen Centre for Cancer and Health, Copenhagen, Nørrebro, Denmark

REFERENCES:
- [Derived] Sommer MS, Trier K, Vibe-Petersen J, Missel M, Christensen M, Larsen KR, Langer SW, Hendriksen C, Clementsen P, Pedersen JH, Langberg H. Perioperative rehabilitation in operation for lung cancer (PROLUCA) - rationale and design. BMC Cancer. 2014 Jun 4;14:404. doi: 10.1186/1471-2407-14-404. PMID 24898680